CLINICAL TRIAL: NCT04712734
Title: An Open-label, Adaptive, Repeat-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Iloperidone Long-acting Injection (LAI) in Patients With Schizophrenia
Brief Title: A Study to Evaluate Iloperidone Long-acting Injection (LAI) for the Treatment of Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VYV-683-1005
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iloperidone (Experimental)
  Interventions: Drug: Iloperidone

INTERVENTIONS:
Drug: Iloperidone — oral tablet, long-acting injection
  Other Names: VYV-683

SUMMARY:
This is a multicenter, open-label, adaptive, repeat-dose study to evaluate the safety, tolerability, and pharmacokinetics of iloperidone long-acting injection (LAI) in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Male or female patients 18 to 65 years of age (inclusive).
* Clinical diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorder (DSM-5) for at least 1 year.
* Symptomatically stable within the past two months.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs.
* Pregnant or nursing (lactating) women.
* A positive test for drugs of abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of iloperidone and its metabolites following repeat-dosing of iloperidone given as a long-acting injection. | 24 weeks
  As measured by plasma concentrations.
Assessment of safety and tolerability of repeat-dosing of iloperidone given as a long-acting injection. | 24 weeks
  As measured by spontaneous reporting of adverse events (AEs).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Vanda Investigational Site, Garden Grove, California
  - Vanda Investigational Site, Gaithersburg, Maryland
  - Vanda Investigational Site, Marlton, New Jersey